CLINICAL TRIAL: NCT04295746
Title: Improving Daily Living Skills in People With Autism Spectrum Disorder Through a Personalised Serious Game
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Ersilia Vallefuoco, PhD, Federico II University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9820
Record Dates: First submitted 2020-02-29; First posted 2020-03-04 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; serious game
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serious Game ShopAut (Experimental): Each participant played 10 game sessions, one per week, for no more than 30 minutes.
  Interventions: Other: Serious Game ShopAut

INTERVENTIONS:
Other: Serious Game ShopAut — The serious game ShopAut, is a three-dimensional game conceptually based on classic 3D life simulation games. ShopAut aims to teach players the procedure of a shopping activity; to reinforce object categorization and recognition in a supermarket; to improve attention, orientation, and problem-solving skills; and to help the player engage in simple economic transactions.
  The intervention provides a virtual training with ShopAut to train, experiment, and practice behaviours and actions that can be then transferred in real-life contexts.

SUMMARY:
This study evaluates the efficacy of a rehabilitation intervention for people with Autism Spectrum Disorder through an individualised serious game developed for improving skills related to a specific daily living activity: shopping in a supermarket.

DETAILED DESCRIPTION:
Serious games are innovative computer-based interventions to support children and adults with Autism Spectrum Disorder (ASD). However, few studies have assessed the efficacy of these interventions in real-life contexts. The present study investigates the generalisation of daily living skills related to shopping activities after a rehabilitation intervention administered via a personalised serious game (ShopAut). The underlying hypothesis of this study is that training with an individualised serious game can improve performance in a real-life environment. In order to prove this hypothesis, a small sample of subjects with ASD will play an individualised serious game, ShopAut, for ten sessions. Subjects will undergo real-life experiences in a supermarket pre- and post-virtual training to determine whether there had been a generalisation of skills from the virtual environment to the real environment. Improvements in skills and performance in the real shopping activity are evaluated using specific tools.

The serious game ShopAut is developed integrating an individualised design that provides both the personalisation of the game's scenario, contents, difficulty, and user interface; and the customisation of game modes, player perspectives, and input devices. It is a three-dimensional game that provides a realistic shopping experience where the player can practice and engage with, above all, shopping activities, experiment their problem-solving skills, and take on unexpected events.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Autism Spectrum Disorder, in keeping with the diagnostic criteria of Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V)
* chronological age between 8 and 16 years
* a rehabilitation plan already underway in accordance with the study's goals
* Representatives of parental authority who gave informed written consent
* native Italian speakers

Exclusion Criteria:

* no physical impairments
* participant to another research protocol
* known organic syndrome and/or non-stabilized neuropediatric (e.g. seizures) or medical (e.g. diabetes mellitus) comorbidities

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
change from baseline in a specific evaluation form based on the International Classification of Functioning, Disability and Health: children and youth version (ICF-CY) at 11 weeks | baseline and 11 weeks
  In order to describe the participants' functioning in the supermarket, an ad hoc evaluation form was created based on the International Classification of Functioning, Disability and Health: children and youth version (ICF-CY). The form follows the ICF-CY scale so higher scores mean a worse outcome.
change from baseline in Vineland Adaptive Behavior Scale II (VABS-II) at 6 months | baseline and 6 months
  The Vineland Adaptive Behavior Scale II (VABS-II) is a standardized paediatric functional assessment tool. The VABS-II offers a way to measure personal and social self-sufficiency in real-life situations and to observe how these cognitive abilities impact the autonomy management process when put into practice. The VABS-II consists in a semi-structured interview with the parents. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Vineland Adaptive Behavior Scale II (VABS-II) at 12 months | 12 months
  The Vineland Adaptive Behavior Scale II (VABS-II) is a standardized paediatric functional assessment tool. The VABS-II offers a way to measure personal and social self-sufficiency in real-life situations and to observe how these cognitive abilities impact the autonomy management process when put into practice. The VABS-II consists in a semi-structured interview with the parents. Higher scores mean a better outcome.
a specific evaluation form based on the International Classification of Functioning, Disability and Health: children and youth version (ICF-CY) at 12 months | 12 months
  In order to describe the participants' functioning in the supermarket, an ad hoc evaluation form was created based on the International Classification of Functioning, Disability and Health: children and youth version (ICF-CY). The form follows the ICF-CY scale so higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Pepino, Study Director — Federico II University
Locations (1):
- University of Naples Federico II - Centro Medico Riabilitativo Pompei, Naples, Italy

IPD SHARING:
Plan to Share IPD: No